CLINICAL TRIAL: NCT05897918
Title: Topical 10% Tranexamic Acid in Treatment of Facial Erythema and Telangiectasia With or Without Microneedling Comparative Study
Brief Title: Tranexamic Acid in Treatment of Facial Erythema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Leila Gallab Mahmoud Mohamed, qena, Al-Azhar University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSc/AZAST/DVA021/18/215/1/2023
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Patient With Facial Erythema
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single group (Other)
  Interventions: Drug: Tranexamic Acid 500 MG

INTERVENTIONS:
Drug: Tranexamic Acid 500 MG — Each patient received treatment on both sides of the face, one side treated by micro needling with 10% topical tranexamic acid, and othert side treated by 10% topical tranexamic acid alone every 2 weeks for 3 sessions

SUMMARY:
Our aim is to evaluate the efficacy of 10% topical tranexamic acid with microneedling in treatment of facial erythema

DETAILED DESCRIPTION:
Facial erythema is redness of the skin or mucous membranes, occurs because of cutaneous blood vessel dilatation and increased blood flow to the skin.it most noticeable in fair-skinned individuals, it may be transient erythema (flushing), persistent erythema, or perilesional erythema around papules and pustules .

Flushing is a transient erythema, usually a physiological phenomenon due to strong emotion, exercise, heat exposure, hyperthermia, spicy food and alcohol intake. But it may be pathological due to pheochromocytoma, carcinoid syndrome .

Persistent erythema is facial erythema that lasts for at least 3 months. It may be due to primary skin diseases such as rosacea, demodicosis, contact dermatitis, polymorphous light eruption, acne, drug-induced (cortisone, brimonidine), lupus erythematosus or due to systemic diseases as mastocytosis, dermatomyositis and hyperthyroidism Rosacea is a chronic inflammatory skin disease characterized by erythema, papules, pustules and telangiectasia affecting the central of the face, women are more often affected than men , there are several theories regarding the cause of rosacea, including genetic, environmental, vascular, and inflammatory factors, rosacea is classified into four main subtypes erythematotelangiectatic, papulopustular, phymatous, and ocular type

Cutaneous lupus erythematosus (LE) is a common autoimmune disease which is limited to the skin, manifested with malar erythema (butterfly eruption),discoid lesions, photosensitivity . It is caused by a complex interplay between genetics, hormones and environmental factors, potential environmental triggers are ultraviolet (UV) radiation and smoking. , histopathologic findings, immunofluorescence, and antinuclear antibodies will aid in making the diagnosis Contact dermatitis of the face can present as a result of a topical causative agent, and it may represent an irritant contact dermatitis, allergic contact dermatitis. A detailed patient history reveals the application of a topical formulation or the contact with a possible precipitating factor will guide the correct diagnosis .

Acne is a multifactorial disorder of the pilosebaceous unit, characterized by non-inflammatory open or closed comedones and inflammatory papules, pustules, and nodules. may present with facial redness typically affects the areas of skin with the highest density of sebaceous follicles including the face, upper chest and back, A cardinal differential diagnosis point is the presence of comedones in acne Drug induced facial erythema due to long term use of a topical corticosteroid or after its abrupt discontinuation after long-term application. It presents with erythema, telangiectasia and papules on the areas of corticosteroid application, diagnosis is based on the monomorphic nature of lesions and the reported history of chronic application of a corticosteroid.

Polymorphous Light Eruption (PLE) is a common photodermatosis characterized by erythematous papules, papulovesicular, and plaques on sun-exposed areas like the face, neck, the eruption appear immediately or several hours after sun exposure and the typical occurrence in spring and early summer .

As not every patient with a facial erythema is the same so, the approach to the patient with a 'red face' includes detailed medical history , whole-body examination and additional laboratory tests are required to confirm the suspected diagnosis .

Traditional options for treatment of facial erythema include the topical brimonidine tartrate , oxymetazoline , have high recurrence rate and Pulsed Dye Laser or Intense pulsed light (IPL) they are rather expensive , although these methods usually show satisfactory results, they are unable to meet the modern patient's need to improve his/her appearance. Therefore, novel and more effective treatment sought by dermatologists.

Tranexamic acid, is an antifibrinolytic drug (synthetic lysine-like molecule) that Works by preventing blood clots from breaking down too quickly , it is used to prevent excessive blood loss from major trauma, postpartum bleeding, heavy menstruation and nose bleeds Tranexamic acid acting by competitively inhibits the activation of plasminogen to plasmin so, suppress plasmin-induced angiogenesis. It also suppressing pro-inflammatory cytokines (interleukin 6 and tumor necrosis factor alpha). Moreover, it can restore the compromised epidermal permeability barrier function and thus decreasing erythema . So, we aimed to evaluate the efficacy of 10% topical tranexamic acid in treatment of facial erythema with microneedling.

ELIGIBILITY:
Inclusion Criteria:

Female Patients clinical diagnosis with persistent facial erythema and telangiectasia. Co-operative patient and patients willing for the procedure

Exclusion Criteria:

active infection at the local site or recurrent herpes. bleeding disorders or anticoagulant medications scar and keloid formation. unrealistic expectations. Pregnant or lactating women

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
change in facial erythema | after 6 week of end point
  method of measurement by clinician erythema assessment score Description Score Clear skin with no signs of erythema 0 Almost clear; slight redness 1 Mild erythema, definite redness 2 Moderate erythema; marked redness 3 Severe erythema; fiery redness 4
  by clinician erythema assesment score

CONTACTS AND LOCATIONS:
Locations (1):
- Azhar University, Asyut, Egypt

REFERENCES:
- See also: Red face revisited: Flushing 2014. — https://doi.org/10.1016/j.clindermatol.2014.02.019
- See also: red face': not always rosacea 2016. — https://doi.org/10.1016/j.clindermatol.2016.10.015
- See also: The Great Mimickers of Rosacea 2014. — https://europepmc.org/article/med/25101343